CLINICAL TRIAL: NCT01541514
Title: Evaluating the Patient-Ventilator Synchrony During Mechanical Ventilation in Patients With Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0172
Record Dates: First submitted 2012-01-17; First posted 2012-03-01 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Mechanically Ventilated ICU Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall purpose to the study is to prospectively study how often patients with and without acute lung injury (ALI) have patient-ventilator asynchrony demonstrated as stacked breaths. The investigators seek to describe the quantity of stacked breaths by continuously recording flow, volume, and pressure waveforms routinely displayed on the vent. The investigators also seek to describe how primary ICU teams manage asynchrony documenting interventions of sedation or vent manipulation and what modality is most successful.

ELIGIBILITY:
Inclusion Criteria:

age > 18 years intubated and mechanically ventilated diagnosed with acute lung injury (ALI) or requiring mechanical ventilation for reasons other than ALI

Exclusion Criteria:

neurological deficits (acute or chronic) that prevent effective diaphragm activity.

* Neuromuscular disease affecting the diaphragm
* Neuromuscular blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult ICU patients receiving mechanical ventilation
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
double stacks | number per minute over 5 minutes
  ventilator waveform recording

SECONDARY OUTCOMES:
level of sedation | baseline
  Richmond Agitation Sedation Score
mode of ventilation | 30min
  ventilator adjustment

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hall, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States